CLINICAL TRIAL: NCT01543100
Title: Prognostic Study of Markers of Angiogenesis and Coagulability in Patients With Monoclonal Gammopathy
Acronym: PACMoG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LOC/10-02 - PACMoG; 2010-A00378-31 (Other: ID RCB); B100413-10 (Other: AFSSAPS); 10/16-758 (Other: CPP Rennes)
Record Dates: First submitted 2011-08-23; First posted 2012-03-02 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Monoclonal Gammopathy; Monoclonal Gammopathy of Undetermined Signification; Myeloma
Keywords: MGUS
MeSH Terms: conditions — Paraproteinemias; Neoplasms, Plasma Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- monoclonal gamopathy (Experimental): Patients with monoclonal gammopathy either MGUS or myeloma at diagnosis or more than 3 months after a first myeloma treatment with chemotherapy and/or antiangiogenic drugs.
  * Patient's age ≥18 yo,
  * Patients having signed the specific consent of the study.
  Interventions: Other: blood and bone marrow samples

INTERVENTIONS:
Other: blood and bone marrow samples — Specific tests of the study will be realized from :
  * Blood samples: 2 EDTA tubes and 1 tube without anticoagulant per included patient.
  * Bone marrow: 3 ml collected during of myelogram punction made for the diagnosis.
  In all cases, no additional sampling will be performed.

SUMMARY:
Blood circulating endothelial cells (CEC) and microparticles (MPs) are described in the literature to be associated with vascular failures and dysfunction that reflect neo-angiogenesis and risk of thrombosis, respectively. There a few number of CEC in healthy patients although they significantly increase in several cancers including myeloma. However, no study explored to date a correlation of CEC and/or circulating endothelial progenitors (CEP) and MPs with the tumoral growth of monoclonal gammopathy. On the other hand, there is no study measuring the CEC and CEP directly in the bone marrow. The investigators aim is to evaluate these 2 original features in patients with monoclonal gammopathy: monoclonal gammopathy of undetermined signification (MGUS) and myeloma. This is a preliminary multicentric study.

DETAILED DESCRIPTION:
Principal objective : Research of a correlation of blood CEC and MPs with the tumoral volume and the clinico-biological staging of monoclonal gammopathies.

Secondary objectives : Research of a correlation of bone marrow endothelial cells and MPs, both measured by flow cytometry, with the tumoral volume and the clinico-biological staging of monoclonal gammopathies.

Principal analyses : Blood levels of CEC and its progenitors, soluble parameters of angiogenesis and of coagulability, and microparticles versus classical indicators of tumoral growth of monoclonal gammopathies (beta2-microglobulin and Ig peak).

Secondary analyses : Bone marrow levels of endothelial cells and its progenitors, soluble parameters of angiogenesis and of coagulability, and microparticles versus classical indicators of tumoral growth of monoclonal gammopathies (beta2-microglobulin and Ig peak).

Methodology : PACMoG is an interventional, prospective and multicentric pilot study. Biologic parameters will be determined at the diagnosis of monoclonal gammopathy. Results will be compared to the monoclonal gammopathy international staging and the clinical follow-up.

Procedures : Specific tests of the study will be realized from :

* Blood samples: 2 EDTA tubes and 1 tube without anticoagulant per included patient.
* Bone marrow: 3 ml collected during of myelogram punction made for the diagnosis.

In all cases, no additional sampling will be performed.

Specific analyses :

- Specific biological assays in blood and bone marrow will be:

* Endothelial and progenitor cells levels
* Number and cellular origin of MPSs
* Levels of phospholipid-dependant coagulability
* Soluble parameters of angiogenesis (VEGF, soluble CD146, endostatin)
* Soluble parameters of coagulability (Levels of thrombomodulin, tissue factor and D-Dimer)

ELIGIBILITY:
Inclusion Criteria:

* Patients with monoclonal gammopathy either MGUS or myeloma at diagnosis or more than 3 months after a first myeloma treatment with chemotherapy and/or antiangiogenic drugs.
* Patient's age ≥ 18 years old,
* Patients having signed the specific consent of the study.

Exclusion Criteria:

* Treatment with chemotherapy and/or antiangiogenic drugs at the inclusion
* Age < 18 years old
* No specific consent of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Blood levels of CEC and its progenitors | Day 1
  Blood levels of CEC and its progenitors
Blood levels of soluble parameters of angiogenesis and of coagulability | Day 1
  Blood levels of soluble parameters of angiogenesis and of coagulability
Blood levels of microparticles versus classical indicators of tumoral growth of monoclonal gammopathies (beta2-microglobulin and Ig peak). | Day 1
  Blood levels of microparticles versus classical indicators of tumoral growth of monoclonal gammopathies (beta2-microglobulin and Ig peak).

SECONDARY OUTCOMES:
Bone marrow levels of endothelial cells and its progenitors | Day 1
  Bone marrow levels of endothelial cells and its progenitors
Bone Marrow levels of soluble parameters of angiogenesis and of coagulability | Day 1
  Bone Marrow levels of soluble parameters of angiogenesis and of coagulability
Bone Marrow levels of microparticles versus classical indicators of tumoral growth of monoclonal gamopathies (beta2-mcicroglobulin and Ig peak). | Day 1
  Bone Marrow levels of microparticles versus classical indicators of tumoral growth of monoclonal gamopathies (beta2-mcicroglobulin and Ig peak).

CONTACTS AND LOCATIONS:
Overall Officials: Benoît GUILLET, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France